CLINICAL TRIAL: NCT07090668
Title: Trans-auricular Nerve Stimulation as an Innovative Approach to the Treatment of Pain in Pediatric Patients Suffering From Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Anna Woodbury, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00008398
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
Keywords: sickle cell disease; pain management in Sickle cell disease; Trans-auricular vagal nerve stimulation; trans-auricular nerve stimulation
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Controlled, single blind feasibility study. Controls will be historical controls, consisting of patients with similar clinical presentations who did not receive tAN
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Controls (Same participant but past data) (No Intervention): Participants will serve as their own controls. Using chart review, we will collect data from each participant's previous admission for a pain crisis during which they did not receive tAN treatment and compare it to their current admission, during which they are being treated with tAN
- tAN group (Experimental): Subjects admitted to CHOA with SCD pain crisis.
  Interventions: Device: tAN device

INTERVENTIONS:
Device: tAN device — Sparrow Link tAN device from Spark Biomedical, a non-invasive, adhesive earpiece placed over branches of the trigeminal nerve and vagus nerve near the tragus and mastoid around the ear. The stimulation level is titrated by the investigator to a perceptible but comfortable intensity. Patients cannot adjust the settings themselves, though adjustments can be made upon request.
  The device consists of a disposable earpiece connected by a cable to a battery-powered controller (3 AAA batteries). It emits a biphasic, rectangular waveform with a 100 µs interphase and a maximum output of 95V.
  Arms: tAN group

SUMMARY:
The goal of this study is to evaluate the effects of transauricular vagus and trigeminal nerve stimulation on the treatment of pain in children with Sickle Cell Disease.

* The primary objective is to determine the feasibility of using a tAN device to treat pain in pediatric participants with SCD by assessing the completion rate, stimulation tolerability, and acceptability of the intervention measures.
* The secondary objective is to assess the preliminary efficacy of using a tAN device as a remedy for pain in pediatric SCD subjects by analyzing inflammatory serum biomarker levels, the Functional Status Scale (FSS), the Wong-Baker FACES questionnaire, tracking analgesic consumption, and other assessments.

DETAILED DESCRIPTION:
The vagus nerve, the body's longest cranial nerve, extends from the brainstem to deep regions of the gastrointestinal tract and plays a vital role in regulating parasympathetic activity across multiple organ systems, including the cardiovascular, respiratory, immune, and nervous systems. Since the early 2000s, vagal nerve stimulation (VNS) has been explored as a therapeutic tool across various diseases, particularly for pain management. VNS can reduce pain by three primary mechanisms: 1) suppressing systemic inflammation, 2) modulating central pain-processing pathways, and 3) alleviating depressive symptoms, which are known to intensify the experience of pain.

Sickle cell disease (SCD) is a genetic blood disorder caused by a point mutation in the β-globin gene, resulting in the production of abnormal hemoglobin (HbS). This leads to polymerization of hemoglobin under low-oxygen conditions, which causes red blood cells to become rigid and sickle-shaped. These malformed cells damage blood vessels and adhere to endothelial surfaces, resulting in vaso-occlusion and impaired blood flow. The subsequent ischemia-reperfusion injury provokes widespread inflammation and produces both acute pain episodes and chronic pain syndromes, often beginning in childhood and persisting throughout life.

The current standard for managing SCD-related pain often involves chronic opioid use, which can lead to dependence, tolerance, and serious side effects. Given the ongoing opioid crisis, there is an urgent need for non-pharmacologic alternatives that are safe, effective, and scalable.

This study proposes the use of transcutaneous auricular vagal nerve stimulation (taVNS) as well as trigeminal auricular nerve stimulation (TAN) -non-invasive methods that stimulates vagal afferents and branches of the trigeminal nerve through the ear-to treat pain in pediatric patients with SCD. taVNS is notable for its excellent safety profile, with minimal to no adverse effects reported in clinical studies. It is a multimodal pain management tool, acting simultaneously on immune, neurologic, and psychological pathways that contribute to pain in SCD.

The innovative aspect of this study lies in its application of a non-invasive, neuroimmune-modulating therapy in a pediatric population with complex pain needs. By potentially reducing the frequency and severity of pain episodes and thereby decreasing reliance on opioids, tAN could transform the clinical approach to pain management in SCD. Ultimately, this research aims to provide a safe, sustainable, and accessible intervention that addresses both the biological and psychosocial dimensions of pain in children and adolescents with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of sickle-cell anemia (HbSS)
* Normal outer ear anatomy and intact skin for tAN placement
* Hospitalized for a pain crisis and experiencing pain as a result of SCD
* Patients must have had at least one prior hospitalization for a sickle cell pain crisis in the past

Exclusion Criteria:

* History of seizures
* History of uncontrolled psychiatric illness
* Repeated episodes of autonomic instability (apnea or bradycardia) that are not self-resolving
* Cardiomyopathy
* Diagnosis of Acute Chest Syndrome
* Unrepaired congenital anomalies affecting the cardiovascular or respiratory system
* Hemodynamically unstable patients
* Females who are pregnant or lactating. Subjects who refuse a pregnancy test.
* Women of childbearing potential, not using adequate contraception as per the investigator's judgment, or not willing to comply with contraception for the duration of the study
* Patients with a history of surgery within the last 3 months
* Patients who suffered from a stroke within the last 3 months
* Patient admitted with a fever or who develops a fever throughout their hospitalization
* Patients whose disease-modifying therapy (HU, chronic transfusions, etc.) and/or pain medications (gabapentin, pregabalin, etc.) have not yet reached a steady dose
* Patients who have had 3 or more hospitalizations for acute pain crises in a given year

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Completion Rate | Through study completion (an average of 3-7 days)
  Completion rate will be calculated by dividing the number of subjects who successfully used tAN for the duration of the trial, divided by the total number of subjects who participated in the trial.
  Subjects who prematurely opt to interrupt their participation in the study will not be included in the cohort of patients who successfully completed the study
Stimulation tolerability | Baseline, everyday throughout the study (an average of 3-7 days)
  Stimulation tolerability will be evaluated daily during hospitalization by asking participants to describe any sensations experienced in response to percutaneous stimulation. Participants will be encouraged to express the sensation in their own words.
  The investigator will then further clarify the nature of the sensation-such as whether it feels like burning, tingling, or stabbing-to better characterize the participant's experience.
Acceptability of intervention | Baseline, everyday throughout the study (an average of 3-7 days)
  Acceptability of intervention measure will be assessed using a standardized 4 item questionnaire.

SECONDARY OUTCOMES:
Wong-Baker FACES | Baseline, everyday throughout the study (an average of 3-7 days)
  The Wong-Baker FACES Pain Rating Scale is a widely used tool to help individuals-especially children-communicate their level of pain. It uses a series of six cartoon faces, ranging from a happy face at 0 ("No Hurt") to a crying face at 10 ("Hurts Worst"), allowing patients to point to the face that best describes their pain.
Functional Status Scale(FSS) | Baseline, everyday throughout the study (an average of 3-7 days)
  The FSS evaluates six functional domains: Mental Status, Sensory Function, Communication, Motor Function, Feeding, Respiratory Status Each domain is scored on a scale from 1 to 5. Total score range: 6 (best possible function) to 30 (worst possible function)
Change in Interleukin 6 (IL-6) levels | Baseline, end of the study (an average of 3-7 days)
  IL-6 is a pro-inflammatory cytokine involved in immune responses, inflammation, and infection.
  Typically < 5 pg/mL in serum or plasma
Change in MCP-1 | Baseline, end of the study (an average of 3-7 days)
  MCP-1 is a pro-inflammatory chemokine that recruits monocytes and other immune cells to sites of inflammation. In children, elevated MCP-1 levels are seen in conditions such as infections, inflammatory diseases Normal levels in healthy children are typically <100-200 pg/mL
Change in Tumor necrosis factor (TNF-α) | Baseline, end of the study (an average of 3-7 days)
  TNF-α (Tumor Necrosis Factor Alpha) is a key pro-inflammatory cytokine involved in immune activation and systemic inflammation.
  Normal levels are typically <10 pg/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Woodbury, MD, Principal Investigator — Emory University
Locations (1):
- Children's Hospital of Atlanta: Eagelston, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No